CLINICAL TRIAL: NCT04144946
Title: Identification of Early Changes in Patellar Tendinopathy Using Ultra-high Field Strength MRI
Acronym: 7TKnee
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Nikolaj Mølkjær Malmgaard-Clausen, Medical Doctor, PhD student, Bispebjerg Hospital
Other Study IDs: BBH-148
Record Dates: First submitted 2019-10-18; First posted 2019-10-30 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Tendon Injuries; Tendinopathy; Patella; Tendinitis
MeSH Terms: conditions — Tendon Injuries; Tendinopathy; Patella Fracture

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Bilateral tendon biopsies
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy control group (CTRL): Sports active individuals with no history of patellar tendinopathy.
- Early tendinopathy group (ET): Sports active individuals with clinical signs of early tendinopathy and debut of symptoms within 90 days.
- Chronic tendinopathy group (CT): Sports active individuals with clinical signs of tendinopathy and duration of symptoms >90 days.

SUMMARY:
This project will investigate patellar tendon tissue (transmission electron microscopy of structure and protein analyses) coupled with magnetic resonance imaging (1.5T and 7T) from persons with i) chronic patellar tendinopathy (CT), ii) the earliest possible signs and symptoms of patellar tendinopathy (ET), and iii) symptom free controls (CTRL)(matched for age and physical activity/sports participation).

The investigators hypothesize that 7T MRI will be able to detect more subtle changes in early tendinopathy as compared to 3T MRI, thereby taking advantage of the increased spatial resolution that can be obtained in MRI with higher field strength. Further the investigator hypothesise that alterations in the tissue will be more pronounced in the CT group compared to ET and healthy controls.

DETAILED DESCRIPTION:
Tendon tissue plays an essential role in transmitting contractile forces to bone to produce movement and is therefore uniquely designed to withstand considerable loads (up to ~8 times body weight) during human locomotion. Yet, repetitive use often results in overuse injuries such as tendinopathies, which is a common clinical condition characterized by pain during activity, localized tenderness upon palpation, swelling of the tendon and impaired performance. Tendinopathy is a sizeable problem in both elite and recreational athletes. In fact, the incidence of tendon injuries has been estimated to be as high as 30-50% of all sports injuries, and 50% of elite endurance runners, and 6% of sedentary people will at some point experience a tendon injury. Moreover, the symptoms and reduction in performance may be quite protracted and last for years. To date the ability to detect the early onset of the disease, and thus to prevent it from becoming chronic and debilitating, remains an enigma and the investigators wish to bridge this gap in knowledge by studying patellar tendon tissue samples coupled with magnetic resonance imaging (3T and 7T)

ELIGIBILITY:
Inclusion Criteria:

Common for all groups

* Sports active individuals.
* Age [18-45] years old.
* BMI [18.5-30]

ET - group

* Symptom onset within 90 days at inclusion
* Clinical signs of patellar tendinopathy.
* Activity related pain in the patellar tendon.
* Palpation pain in the proximal part of the patellar tendon.
* At least one of the following three changes on the ultrasound scanning:

  * Thickening of the AP diameter on the symptomatic side.
  * Increased Power Doppler signal on the symptomatic side.
  * Hypoechogenic area corresponding to the symptomatic area of the tendon.

CT - group,

* Symptom onset >90 days ago
* Clinical signs of patellar tendinopathy.
* Activity related pain in the patellar tendon.
* Palpation pain in the proximal part of the patellar tendon.
* At least one of the following three changes on the ultrasound scanning:

  * Thickening of the AP diameter on the symptomatic side.
  * Increased Power Doppler signal on the symptomatic side.
  * Hypoechogenic area corresponding to the symptomatic area of the tendon.

CTRL - group - Similar activity level as the two patient groups.

Exclusion Criteria:

Common for all groups

* Previous surgery in the knee on the ipsilateral side.
* Previous corticosteroid injection in the patellar tendon on the ipsilateral side.
* Smoking
* Known arthritis
* Known diabetes
* Known hypercholesterolemia
* Previous injections in the ipsilateral tendon.
* MRI contraindications

  * Ferromagnetic objects
  * Pregnancy
  * Lactation

ET - group

* Previous injuries in the patellar tendon on the ipsilateral side.
* Started systematized treatment.

CTRL - group

- Previous injuries in the patellar tendon on the ipsilateral side.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Sports active individuals
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2019-10-18 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Cross sectional area (CSA) on Magnetic Resonance Imaging knee scans | 0 months, observational cross sectional study.
  Magnetic Resonance Imaging of the knee, used to measure cross sectional area (cm^2)
Decay times from Magnetic Resonance Imaging knee scans | 0 months, observational cross sectional study.
  Magnetic Resonance Imaging of the knee used to calculate decay times (ms) in the tendon tissue.
Patellar tendon biopsies | 0 months, observational cross sectional study.
  Tendon biopsies obtained with bard magnum instrument approximately 10 mg. Used for quantitative mRNA measures expressed as relative values to the expression of a housekeeping gene with stable expression (AU).

SECONDARY OUTCOMES:
International Physical Activity Questionnaire (IPAQ) | 0 months, observational cros sectional study.
  IPAQ categorical scores (High, moderate or low activity level) will be reported, to characterise participants activity level
Body Mass Index | 0 months, observational cross sectional study.
  BMI
Questionnaires - weekly activity level (time consumption) | 0 months, observational cross sectional study.
  hours/week spend on leisure time activities loading the legs.
Questionnaires - Numerical Rating Scale (NRS) - Pain | 0 months, observational cross sectional study.
  range 0-10, 10 being the highest possible pain level and 0 being no pain.
VISA-P | 0 months, observational cross sectional study.
  Standardised score of functional capability, in patient with patellar tendinopathy. Total score will be reported; scale (0-100). 100=full functional capacity 0=poor functional capacity.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kjær, Professor, Principal Investigator — Institute of Sports Medicine, Copenhagen
Locations (1):
- Institute of Sports Medicine Copenhagen, Copenhagen, NV, Denmark

IPD SHARING:
Plan to Share IPD: Undecided